CLINICAL TRIAL: NCT04713761
Title: Clinical Study of Neoadjuvant Anti-PD-1 Drug Toripalimab Combined With Chemotherapy in the Treatment of Locally Advanced Epithelial or Mixed Tissue Malignant Pleural Mesothelioma
Brief Title: Neoadjuvant Toripalimab Combined With Chemotherapy in the Treatment of Malignant Pleural Mesothelioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Director of thoracic department, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-010(FK-NEO-MPM-001)
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Malignant Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — toripalimab; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab (Experimental)
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Neoadjuvant treatment stage: Toripalimab 240mg, Carboplatin AUC5+ pemetrexed 500 mg/m ², iv, 3 weeks per cycle, 2-4 cycles in total; Surgical treatment stage: Patients with MPM received surgical treatment (PD/EPP) after neoadjuvant therapy. Patients who were unable to operate or refused surgical treatment due to various reasons were treated with multidisciplinary discussion.
  Adjuvant treatment stage: CR, PR and SD patients who have been treated surgically: Toripalimab 240mg, Carboplatin AUC5+ pemetrexed 500 mg/m ²,iv, up to 4 cycles (including neoadjuvant stage).
  Other Names: carboplatin; pemetrexed

SUMMARY:
This is a single-arm, open, II phase study to evaluate the safety and efficacy of Toripalimab, pemetrexed and carboplatin in the treatment of locally advanced malignant MPM in 15 newly diagnosed patients with locally advanced malignant MPM.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent;
* Age ≥ 18 years;
* Histology or cytology confirmed upper or mixed type of MPM, and previously untreated;
* Imaging confirmed that MPM was locally advanced;
* PET-CT confirmed no metastasis;
* ECOG physical status score 0-1;
* Life expectancy at least 12 weeks.
* Have measurable lesions
* Good function of other major organs (liver, kidney, blood system, etc.):-absolute neutrophil count ((ANC) ≥ 1.5 × 109), platelet (≥ 100 × 109), hemoglobin (≥ 90g/L). Note: patients shall not receive blood transfusion or growth factor support within 14 days before blood collection during the screening period;-International standardized ratio (INR) or prothrombin time (PT) ≤ 1.5 × normal upper limit (ULN);-activated partial thromboplastin time (APTT) ≤ 1.5 × ULN;- serum total bilirubin ≤ 1.5 × ULN (Gilbert syndrome patients with total bilirubin must be < 3×ULN). Fertile female patients with aspartate and alanine aminotransferase (AST and ALT) ≤ 2.5 × ULN, or liver metastasis with AST and ALT ≤ 5 × ULN
* Fertile female patients must voluntarily take effective contraceptive measures more than 120 days after chemotherapy or the last administration of triplizumab, whichever is later, and the urine or serum pregnancy test results less than 7 days before entering the group were negative.
* Unsterilized male patients must voluntarily take effective contraceptive measures ≥ 120 days after chemotherapy or the last administration of triplizumab, whichever is the later.

Exclusion Criteria:

* Any systemic anticancer therapy for MPM, including surgery, local radiotherapy, cytotoxic drug therapy, targeted drug therapy and experimental therapy;
* Any Chinese herbal medicine used to control cancer was used within 14 days before the first administration of the study drug;
* Patients with malignant tumors other than MPM in the five years before the start of this trial.
* Complicated with unstable systemic diseases such as uncontrolled hypertension, severe arrhythmias, etc.;
* Active, known or suspected autoimmune diseases, or autoimmune paraneoplastic syndrome requiring systemic treatment;
* Allergic to experimental drugs;
* Previous or current interstitial lung disease;
* Complicated with HIV infection or active hepatitis.
* Those who were injected with vaccines or antibiotics within 4 weeks before the start of this trial, or who had undergone other major operations or severe injuries within the previous 2 months;
* Clinically uncontrolled pleural effusion or ascites requiring pleural or abdominal puncture drainage within 2 weeks before admission;
* Pregnant or lactating women;
* Any malabsorption;
* Those with neurological diseases or mental disorders.
* Participated in another therapeutic clinical study at the same time;
* Other researchers did not consider it appropriate to enroll in the group.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response (MPR) | up to 4 months
  MPR is defined as the proportion of participants who have achieved major pathologic response (on routine hematoxylin and eosin staining, tumors with no more than 10% viable tumor cells) in all participants who have completed the neoadjuvant therapy before surgery.
Health related quality of life (HRQol) | up to 6 months
  The assessment is made according to the Quality of Life Scale for Lung Cancer Patients (EORTC-QLQ-C30 & LC13, Version 3). EORTC's QLQ-C30 & LC13 (V3.0) is a core scale for lung cancer patients, with a total of 43 items. Among them, Item 29 and 30 are divided into seven grades, which are assigned with 1 to 7 scores according to the answer options. The other items are divided into 4 grades: No
Safety: frequency of severe adverse events | up to 5 months
  The frequency of severe adverse events from the participants enrolling to 30 days after the last drug administration or 30 days after surgery or new anti-cancer therapy, which comes first.

SECONDARY OUTCOMES:
Overall survival (OS) | up to 60 months
  It is defined as the time from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date. In the event of a patient with the survival status unknown, the date when the patient is last known to be alive will be used for interpolation (censoring).
Duration of remission (DOR) | up to 60 months
  According to the time from the first recording of objective remission to relapse or death from any cause determined by RECISTv1.1, whichever occurs first.
Disease control rate (DCR) | up to 60 months
  The proportion of patients whose best overall remission (BOR) is CR, PR or disease stable (SD) according to RECISTv1.1 evaluation
Progression-free survival (PFS) | up to 60 months
  PFS is defined as the time from the enrollment of the subject to the first determination of disease progression or death of any cause according to RECISTv1.1, whichever occurs first.

IPD SHARING:
Plan to Share IPD: Undecided